CLINICAL TRIAL: NCT04522726
Title: Clinical Exploring Study of Weiyang Yuping Decoction in Preventing Acute Attacks of Mild to Moderate Intermittent Asthma Based on the Theory of "Preventing Disease From Exacerbating" in Chinese Medicine
Brief Title: A Clinical Study on the Prevention of Mild to Moderate Intermittent Asthma With Chinese Medicine Weiyang Yuping Fang
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020LHSB022
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-03

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma; Traditional Chinese Medicine
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: One group was given Weiyang Yupingfang Granules orally for 1 month on the "Sanfu"days and on the "Sanjiu" days each year for a total of 2 months one year; the other group was given Weiyang Yupingfang Granules orally for 1 month in the first month of each quarter in the four quarters of the year, for a total of 4 months one year.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Treatment group A received Weiyang Yupingfang Granules orally for 1 month on the "Sanfu" days and on the"Sanjiu"days each year for a total of 2 months a year.
  Interventions: Drug: Weiyang Yuping Fang
- Treatment group B (Experimental): Treatment group A received Weiyang Yupingfang Granules orally for 1 month in the first month of each quarter in the four quarters of the year, for a total of 4 months a year.
  Interventions: Drug: Weiyang Yuping Fang

INTERVENTIONS:
Drug: Weiyang Yuping Fang — Weiyang Yuping fang is a combination of the classic ancient Yuping dispersion used to prevent qi deficiency and susceptibility and Bushen Naqi granules optimized formated by Professor Shao Changrong's experience in treating chronic cough and asthma.
  Other Names: Weiyang Yuping granules

SUMMARY:
Clinical exploring study of Weiyang Yuping Decoction in preventing acute attacks of mild to moderate intermittent asthma Based on the theory of "Preventing disease from exacerbating" in Chinese medicine.

DETAILED DESCRIPTION:
Based on the preliminary clinical and basic research, this project intends to highly optimize and integrate the TCM treatment of disease theory with the current methods to form two preventive treatment plans, one treatment group was given Weiyang Yupingfang Granules orally for 1 month on the "Sanfu"days and on the "Sanjiu" days each year for a total of 2 months one year; the other treatment group was given Weiyang Yupingfang Granules orally for 1 month in the first month of each quarter in the four quarters of the year, for a total of 4 months one year.; Comparing the effect of prevention and treatment of mild to moderate intermittent asthma exacerbations of the two prevention methods , provides new ideas for the prevention and treatment of bronchial asthma in the future, and further improves bronchial The level of prevention and treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma according to GINA criteria with a documented history of at least 3 years prior to Visit 1
* Patients have asthma exacerbations every year
* Meet the diagnostic criteria for mild to moderate asthma
* Able to measure lung ventilation function according to ATS (American Thoracic Society) standards
* Patients who have given written informed consent

Exclusion Criteria:

* Medical history of life-threatening asthma including intubation and intensive care unit admission
* Any significant disease or disorder (e.g., cardiovascular, pulmonary other than asthma, gastrointestinal, hepatic, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study
* Pregnancy, breast-feeding or planned pregnancy during the study.
* Participation in another clinical study or took other research drugs during the last 30 days prior to Visit 1
* Known or suspected hypersensitivity to study drugs or excipient
* Suspected poor capability, as judged by the investigator, of following instructions of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Annual severe asthma exacerbation rate | up to 12 months after treatment
  Measured the change from Baseline of annual severe asthma exacerbation rate

SECONDARY OUTCOMES:
Time to first severe asthma exacerbation | up to 12 months after treatment
  Record the time of the patient's first severe asthma exacerbation after treatment
Average change from baseline in pre-dose FEV1 | up to 24 months
  Measured the change from Baseline of forced expiratory volume in the first second
Average change from baseline in pre-dose PEF | up to 24 months
  Measured the change from Baseline of peak expiratory flow
Average change from baseline in Asthma Control Questionnaire | up to 12 months after treatment
  Measured the change from Baseline of Asthma Control Questionnaire (5-item version) - ACQ-5 score

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhui Lu, Doctor, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital Affiliated Shanghai University of TCM, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No